CLINICAL TRIAL: NCT07355894
Title: Health Enhanced Artery Risk Tracking With Widespread Implementation and Screening Effort in AtheroSclerotic CardioVascular Disease (HEARTWISE-ASCVD) Study
Brief Title: Health Enhanced Artery Risk Tracking With Widespread Implementation and Screening Effort in ASCVD (HEARTWISE-ASCVD)
Acronym: HEARTWISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Amgen (Industry); Baylor Scott and White Health (Other); Kaiser Permanente (Other); Vanderbilt University Medical Center (Other); Duke University (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Fatima Rodriguez, Associate Professor of Medicine (Cardiovascular Medicine), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 84062
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Atherosclerotic Cardiovascular Disease (ASCVD); Coronary Artery Calcification
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Notification (Experimental): For participants randomized to notification, the affiliated clinician will receive a message notifying them of the presence of CAC. The notification will include a description of the significance of CAC, provide guideline recommendations, and include a personalized CAC image (as possible). The message will recommend having a risk discussion with the participant. Based on site-level stakeholder feedback, this alert can be retriggered at 2 months for participants who do not have LLT initiation or intensification or LDL-C testing.
  Participants will also receive a notification. Based on stakeholder input, this notification can be delivered centrally or from individual clinicians. The notification will include a description of the significance of CAC, a personalized image (as possible), and recommend a risk discussion with their clinician.
  Interventions: Other: AI-Detected CAC Notification and Care Facilitation
- Delayed Notification (No Intervention): Participants will have their CT scans interpreted and reported according to standard clinical practice. This may mention the presence of CAC in the official radiology imaging report, per usual practice. Participants will not receive any notification beyond this standard of care during the 6-month study period.
  The study team will send a similar notification as the early notification arm to the participants after completion of the study's primary endpoint assessment.

INTERVENTIONS:
Other: AI-Detected CAC Notification and Care Facilitation — After randomization to the early notification arm, the study team will send a standardized notification message to the participant's affiliated clinician. The study team will send a message to the participant after a brief delay. Each site will determine the timing between the initial message to the clinician and the participant based on stakeholder feedback.
  The notification is about the AI-CAC identified on the participant's previous chest CT. It will provide an overview of AI-CAC, a personalized image of AI-CAC, and a recommended risk discussion with their clinician. These clinicians will also be notified of the findings.
  For participants randomized to early notification who do not undergo LLT initiation, intensification, or LDL testing within 2 months, the clinician and participant will receive a second message at that time.
  The participants in the delayed notification arm will receive a similar notification 6 months later.
  Arms: Early Notification

SUMMARY:
This multi-site study will test whether an opportunistic AI-based CAC screening and notification intervention can improve cholesterol treatment and lower cholesterol levels in adults. The study uses artificial intelligence to detect calcium buildup in heart arteries (coronary artery calcium or CAC) on chest CT scans that patients have already had for other reasons. The study will focus on adults who either have known atherosclerotic cardiovascular disease (ASCVD) or have significant calcium buildup (a CAC score of 100 or higher), and whose cholesterol is not well controlled.

It will also evaluate how well this approach can be implemented at scale across multiple health systems. The main questions it aims to answer are:

Does notifying patients and their clinicians about incidental CAC increase lipid-lowering therapy(LLT) initiation or intensification?

Does the intervention improve Low-Density Lipoprotein(LDL)-cholesterol control and related lipid testing?

How does the intervention affect downstream care (e.g., clinic visits, cardiology referrals, and cardiac testing)?

Researchers will use an FDA-cleared AI algorithm to quantify CAC on previously performed non-gated chest CT scans and identify eligible participants through the electronic health record. Participants will be randomized to receive CAC notification either right away or after a 6-month delay.

ELIGIBILITY:
Inclusion Criteria:

* Non-gated chest CT performed within the prior 2 years within the health system
* Active health system engagement with an affiliated clinician eligible for notification, defined as ≥1 clinical visit within the prior 2 years AND at least one of the following:

  1. Active enrollment in the site's integrated healthcare plan (e.g., Kaiser Permanente Northern California), OR
  2. LDL-C measured within the health system within the prior 2 years, OR
  3. Outpatient cardiovascular medication prescription within the prior year
* Meets one of the following clinical criteria:

  1. Clinical ASCVD diagnosis (coronary artery disease, peripheral arterial disease, or ischemic cerebrovascular disease) AND AI-detected CAC >0 on non-gated chest CT, OR
  2. No ASCVD diagnosis AND AI-detected CAC ≥100
* Suboptimal LDL-C control, defined as either: Last LDL-C ≥70 mg/dL in the last 2 years, OR No LDL-C measurement in the last 2 years

Note: Site-level variations and additional refinements may occur based on local stakeholder input and patient population identification.

Exclusion Criteria:

* Dementia
* Heart transplant
* Active hospice
* Other life-limiting illness as determined by the site investigator (e.g., metastatic cancer)
* Additional participant-level exclusions as determined by clinical stakeholders at each site

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120000 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Lipid-lowering therapy initiation or intensification (LLTI) | 6 months after participant randomization
  * Number of new statin prescriptions
  * Number of statin doses/intensity increase
  * Number of PSCK9 inhibitor initiation (monoclonal antibodies and siRNA)
  * Number of Ezetimibe initiations
  * Number of Bempedoic acid initiations

SECONDARY OUTCOMES:
Aspirin prescription | 6 months after participant randomization
  Number of new Aspirin or other antiplatelet prescription
Lipid panel (total cholesterol, HDL-C, LDL-C, triglycerides) ordering | 6 months after participant randomization
  Number of Lipid panel ordering
Lipoprotein(a) test ordering | 6 months after participant randomization
  Number of Lipoprotein(a) test ordering
Changes of total cholesterol, HDL-C, LDL-C, triglycerides, Lipoprotein(a) levels | 6 months after participant randomization
  This outcome measure the changes of the test levels
Healthcare resource use | Baseline through Month 6
  * Number of primary care clinical encounters
  * Number of cardiology encounters
  * Number of coronary artery disease-related imaging tests (e.g. noninvasive stress tests, coronary computed tomography angiography (CCTAs), and angiograms)

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Rodriguez, MD, MPH, Principal Investigator — Stanford University
Locations (6):
- United States (6):
  - University of California, Los Angeles, Los Angeles, California
  - Kaiser Permanente Northern California, Pleasanton, California
  - Stanford University, Stanford, California
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott & White, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No